CLINICAL TRIAL: NCT06346158
Title: Prediction of Propofol Effect-Site Concentration Associated With Deep Anesthesia During Induction of General Anesthesia Based on Electroencephalographic Features: a Prospective Observational Study
Brief Title: Prediction of Propofol Effect-Site Concentration Associated With Deep Anesthesia
Acronym: PRESCOD-AI
Status: Recruiting | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-3615
Record Dates: First submitted 2024-03-08; First posted 2024-04-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia
Keywords: general anesthesia; propofol; interindividual variability; prediction; cognitive performance; electroencephalogram
MeSH Terms: interventions — Electroencephalography; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Cognitive testing — Preoperative cognitive battery test
Device: electroencephalogram — Preoperative 24 channel EEG
Device: High density electroencephalogram — preoperative 128-channel electroencephalogram
Procedure: General anesthesia — induction of general anesthesia using propofol 1%

SUMMARY:
The goal of this observational study is to explore the variability of the concentration at the effect site (Ce) of propofol to reach deep anesthesia (DA) during induction of general anesthesia in adults.

The investigators hypothesized that there is a great variability in this Ce that could be precisely explained by

* Electroencephalographic (EEG) features available prior to induction of anesthesia
* Cognitive performance
* Patients characteristics Participants will undergo preoperative cognitive testing and awake EEG. Then, induction of general anesthesia will be performed using continuous infusion of propofol. The Ce at which Deep anesthesia is observed will be recorded.

DETAILED DESCRIPTION:
Propofol is the most widely used anesthetic to induce general anesthesia (GA). However, as opposed to volatile anesthesia, propofol concentration monitoring is not directly available in humans. Thus, the use of a pharmacokinetic/pharmacodynamic (PK/PD) model in target-controlled infusion (TCI) is recommended. During infusion, the concentration at effect-site (Ce) is assumed to correlate with the level of hypnosis. However, There is a large variability in propofol requirements in common practice. The variability in propofol requirements is attributed to demographic factors, genetic polymorphism, procedure-related changes, and individual sensitivity. Previous studies have shown that EEG characteristics change with age and cognitive status.

Hypothesis : There is a large interindividual variability in patients' sensitivity to propofol which can be precisely modeled using clinical, demographic, and electroencephalographic (EEG) features available prior to induction of general anesthesia. The investigators also hypothesise that this sensitivity to propofol may identify vulnerable brain phenotype related to poor cognitive performance.

Specific objectives: Primary: to investigate the variability of Ce propofol at which deep anesthesia (DA) occurs during induction of general anesthesia (CeDA). Secondary: to explore the relationship between demographics, cognitive performance, and EEG variables with the independent CeDA variable. Tertiary: to develop and validate a machine learning algorithm to predict CeDA based on clinical, demographic and EEG features obtained prior the induction of general anesthesia.

Methods: This prospective monocentric observational study will include 110 participants of 18 years of age or older scheduled for surgery under general anesthesia. Baseline cognitive performance will be assessed using the Montreal Cognitive Assessment. Induction of GA will be performed using 300ml.h-1 of 1% propofol until DA (Defined as a Patient State Index (PSI) < 30) is observed. The primary endpoint will be the Ce propofol at which deep anesthesia (CeDA) occurs as calculated by the Eleveld PK/PD model for propofol. Preoperative raw EEG waveforms from the SedLine monitor will be used to extract statistical, entropic, and spectral features. High-density EEG (128 channels) will also be recorded in a subsample of 40 patients to extract brain functional connectivity features. These features will be entered in a generalized additive model to predict CeDA. We will also develop and validate a machine learning algorithm to predict CeDA based on these features.

Significance/Importance: The results of this study could provide a better understanding of the determinants of the inter-individual variability observed in the pharmacodynamic effect of anesthetic agents. Moreover, the prediction of CeDA may help clinicians in setting the right and safe target in target-controlled infusion of propofol during induction of general anesthesia and further limit the occurrence of deep anesthesia during surgery. Finally, the knowledge of the link between EEG characteristics, sensitivity to anesthetics and cognitive performance may lead to more personalized anesthesia delivery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for any kind of surgery under general anesthesia.
* Adults

Exclusion Criteria:

* Inability to communicate in French or English,
* Known allergy or intolerance or other medical condition that precludes the use of prescribed general anesthesia protocol for this study,
* Patients requiring rapid sequence induction,
* Anticipated or known difficult intubation patient,
* Anticipated or known difficult ventilation patient,
* Body mass index ≥ 35 kg.m-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults' patients scheduled for any kind of surgery in our institution
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Concentration at the effect-site propofol associated with deep anesthesia (CeDA) | during surgery
  Concentration at the effect-site propofol as calculated by the Eleveld model required to reach a Bispectral index < 45 during induction of general anesthesia in micrograms per mL.

SECONDARY OUTCOMES:
Coefficient of determination between statistical, spectral, entropic features extracted from the electroencephalogram and the Concentration at the effect-site propofol associated with deep anesthesia | during surgery
Coefficient of determination between multivariable model and the Concentration at the effect-site propofol associated with deep anesthesia | during surgery
  A generalized additive model will be constructed based on features associated with the Concentration at the effect-site propofol associated with deep anesthesia
Mean absolute error between predicted Concentration at the effect-site propofol associated with deep anesthesia by the machine-learning model and observed Concentration at the effect-site propofol associated with deep anesthesia. | during surgery
  We will developp a machine learning model to predict the Concentration at the effect-site propofol associated with deep anesthesia on a separate database and validate the model on the patients of the present study

OTHER OUTCOMES:
Concentration at the effect-site propofol associated with loss of consciousness (CeLOC) | during surgery
  Concentration at the effect-site propofol as calculated by the Eleveld model required for loss of consciousness during induction of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Louis Morisson, MD, MSc, Principal Investigator — CIUSSS de l'Est de l'Ile de Montréal
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No